CLINICAL TRIAL: NCT07158892
Title: Confirmation of Values and Preferences When Considering a Musculoskeletal Diagnostic Test: A Scenario-Based Study
Brief Title: Understanding Patient Preferences When Deciding on a Voluntary Musculoskeletal Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Associate Dean for Comprehensive Care; Professor and Associate Chair for Faculty Academic Affairs, Department of Surgery and Perioperative Care; Courtesy Professor of Psychiatry and Behavioral Sciences, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004831(2)
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Non-traumatic Musculoskeletal Conditions; Carpal Tunnel Syndrome (CTS); Lateral Epicondylitis; Osteoarthritis; Trigger Digit; Dupuytren Contracture; Rotator Cuff Tendinopathy; De Quervain Disease
Keywords: Musculoskeletal disorders; Diagnostic imaging; Shared decision making; Advance care planning (ACP); Patient preferences; Health communication; Decision conflict; Scenario-Based Study; Orthopedic care
MeSH Terms: conditions — Carpal Tunnel Syndrome; Tennis Elbow; Osteoarthritis; Trigger Finger Disorder; Dupuytren Contracture; De Quervain Disease; Musculoskeletal Diseases; Patient Preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Group 1) (Experimental): Participants randomized to the intervention group will engage in a structured, scenario-based conversation simulating a diagnostic decision-making discussion. This conversation will be guided by a trained researcher using branching scripted prompts designed to reflect an Advance Care Planning (ACP)-style approach. The discussion will explore the participant's values, goals, and understanding of potential benefits and harms of the proposed hypothetical imaging test. No actual diagnostic tests will be ordered.
  Interventions: Behavioral: Diagnostic Advance Care Planning Discussion
- Control (Group 2) (Active Comparator): Participants randomized to the control group will receive the same hypothetical clinical scenario, including mention of a proposed diagnostic imaging test. Instead of a structured discussion, they will be presented with a brief, standardized informational statement describing what the test involves, what it may show, and general risks or limitations. No values-based discussion or simulated conversation will occur.
  Interventions: Behavioral: Informational Statement Only

INTERVENTIONS:
Behavioral: Diagnostic Advance Care Planning Discussion — The intervention consists of a structured, values-based conversation modeled after Advance Care Planning (ACP) principles, adapted for diagnostic decision-making. Participants will receive a hypothetical clinical vignette involving a musculoskeletal diagnostic test (e.g., MRI, X-ray, CT, or ultrasound), followed by a simulated discussion facilitated by a trained researcher. The conversation is guided by branching scripted prompts designed to elicit the participant's values, goals, expectations, and understanding of the potential benefits and harms of testing. Responses are transcribed using verbal-to-text technology. Unlike standard decision aids or educational materials, this intervention emphasizes patient reflection and shared decision-making by prompting participants to consider what matters most to them before making a decision about the test. The discussion does not involve actual test ordering or clinical decisions but is intended to simulate a real-world ACP discussion process.
  Other Names: ACP-style discussion
  Arms: Intervention (Group 1)
Behavioral: Informational Statement Only — Participants will be presented with a brief, standardized informational statement describing what the test involves, what it may show, and general risks or limitations. No individualized values-based discussion or simulated conversation will occur.
  Other Names: Control
  Arms: Control (Group 2)

SUMMARY:
The goal of this clinical trial is to understand how people make decisions about imaging tests for common musculoskeletal problems (like arthritis, tendon problems, or nerve compression). The study involves adult patients attending a musculoskeletal specialty clinic.

The main questions it aims to answer are:

1. Does having a structured conversation about the pros and cons of a test affect how much a person wants to have that test?
2. Does that conversation help people feel more confident and less conflicted about their decision?

Researchers will compare patients who have a values-based discussion with a researcher to those who receive brief written information about the test, to see if these approaches affect how people feel about having the test.

Participants will:

* Read a brief scenario about a proposed diagnostic imaging test (like an X-ray, MRI, CT, or ultrasound).
* Either take part in a short structured conversation or read brief information about the test.
* Answer a short survey about their thoughts on the test.

This study does not involve actual medical testing or affect your clinical care. It is for research purposes only.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years)
* English literacy
* Seeking musculoskeletal specialty care
* Diagnosis of non-traumatic musculoskeletal condition (including but not limited to: carpal tunnel syndrome, lateral epicondylitis, osteoarthritis, trigger digit, Dupuytren's, De Quervain, or rotator cuff tendinopathy)

Exclusion Criteria:

* Cognitive or physical impairment or severe psychiatric illness that would interfere with participation in the scenario-based discussion or completion of the survey instruments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Enthusiasm for proposed hypothetical diagnostic test | Measured using survey on tablet immediately following intervention/control (i.e., ACP-style discussion [Group 1] or informational statement [Group 2])
  Measured using 11-point Likert scale: 0=I would definitely decline this test, 5=I am not sure if I would accept this test, 10=I would definitely proceed with this test.

SECONDARY OUTCOMES:
Decisional conflict regarding the diagnostic test | Measured using survey on tablet immediately following intervention/control (i.e., ACP-style discussion [Group 1] or informational statement [Group 2])
  Assessed using the validated 'SURE' scale (0-4 score; higher scores indicate greater certainty and lower decisional conflict). Please refer to Appendix 2 of PDF study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, Principal Investigator — Dell Medical School, University of Texas at Austin, TX, United States
Locations (1):
- Musculoskeletal Institute, UT Health Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slade SC, Molloy E, Keating JL. 'Listen to me, tell me': a qualitative study of partnership in care for people with non-specific chronic low back pain. Clin Rehabil. 2009 Mar;23(3):270-80. doi: 10.1177/0269215508100468. PMID 19218301
- [Background] Rossettini G, Latini TM, Palese A, Jack SM, Ristori D, Gonzatto S, Testa M. Determinants of patient satisfaction in outpatient musculoskeletal physiotherapy: a systematic, qualitative meta-summary, and meta-synthesis. Disabil Rehabil. 2020 Feb;42(4):460-472. doi: 10.1080/09638288.2018.1501102. Epub 2018 Nov 14. PMID 30428722
- [Background] Rogers CJ, Hackney ME, Zubkoff L, Echt KV. The use of patient-led goal setting in the intervention of chronic low back pain in adults: a narrative review. Pain Manag. 2022 Jul;12(5):653-664. doi: 10.2217/pmt-2021-0118. Epub 2022 Mar 30. PMID 35350847
- [Background] Stellman S, Ellis B, Dawson H, Kocsis A, Mundra J, Hill C, Sahota K, Douglas S. Piloting a new model of personalised care for people with fibromyalgia in primary care with secondary care multidisciplinary support. Musculoskeletal Care. 2023 Jun;21(2):582-591. doi: 10.1002/msc.1708. Epub 2022 Nov 9. PMID 36349698
- [Background] Schenker Y, White DB, Arnold RM. What should be the goal of advance care planning? JAMA Intern Med. 2014 Jul;174(7):1093-4. doi: 10.1001/jamainternmed.2014.1887. No abstract available. PMID 24861458
- [Background] Krones T, Anderson S, Borenko C, Fromme E, Gotze K, Lasmarias C, Lin CP, Neves Forte D, Ng R, Simon J, Sinclair C. Editorial: Advance Care Planning as Key to Person Centered Care: Evidence and Experiences, Programmes and Perspectives. Z Evid Fortbild Qual Gesundhwes. 2023 Aug;180:1-6. doi: 10.1016/j.zefq.2023.07.001. Epub 2023 Jul 26. No abstract available. PMID 37500354
- [Background] van Bokhoven MA, Koch H, van der Weijden T, Grol RP, Kester AD, Rinkens PE, Bindels PJ, Dinant GJ. Influence of watchful waiting on satisfaction and anxiety among patients seeking care for unexplained complaints. Ann Fam Med. 2009 Mar-Apr;7(2):112-20. doi: 10.1370/afm.958. PMID 19273865
- [Background] van Ravesteijn H, van Dijk I, Darmon D, van de Laar F, Lucassen P, Olde Hartman T, van Weel C, Speckens A. The reassuring value of diagnostic tests: a systematic review. Patient Educ Couns. 2012 Jan;86(1):3-8. doi: 10.1016/j.pec.2011.02.003. Epub 2011 Mar 6. PMID 21382687
- [Background] McDonald IG, Daly J, Jelinek VM, Panetta F, Gutman JM. Opening Pandora's box: the unpredictability of reassurance by a normal test result. BMJ. 1996 Aug 10;313(7053):329-32. doi: 10.1136/bmj.313.7053.329. PMID 8760739
- [Background] Kravitz RL, Bell RA, Azari R, Kelly-Reif S, Krupat E, Thom DH. Direct observation of requests for clinical services in office practice: what do patients want and do they get it? Arch Intern Med. 2003 Jul 28;163(14):1673-81. doi: 10.1001/archinte.163.14.1673. PMID 12885682
- [Background] van der Weijden T, van Velsen M, Dinant GJ, van Hasselt CM, Grol R. Unexplained complaints in general practice: prevalence, patients' expectations, and professionals' test-ordering behavior. Med Decis Making. 2003 May-Jun;23(3):226-31. doi: 10.1177/0272989X03023003004. PMID 12809320
- [Background] Epstein RM, Franks P, Shields CG, Meldrum SC, Miller KN, Campbell TL, Fiscella K. Patient-centered communication and diagnostic testing. Ann Fam Med. 2005 Sep-Oct;3(5):415-21. doi: 10.1370/afm.348. PMID 16189057
- [Background] Bedson J, Jordan K, Croft P. How do GPs use x rays to manage chronic knee pain in the elderly? A case study. Ann Rheum Dis. 2003 May;62(5):450-4. doi: 10.1136/ard.62.5.450. PMID 12695159
- [Background] Graham B. The value added by electrodiagnostic testing in the diagnosis of carpal tunnel syndrome. J Bone Joint Surg Am. 2008 Dec;90(12):2587-93. doi: 10.2106/JBJS.G.01362. PMID 19047703
- [Background] Herrle SR, Corbett EC Jr, Fagan MJ, Moore CG, Elnicki DM. Bayes' theorem and the physical examination: probability assessment and diagnostic decision making. Acad Med. 2011 May;86(5):618-27. doi: 10.1097/ACM.0b013e318212eb00. PMID 21436660
- [Background] Karel YH, Verkerk K, Endenburg S, Metselaar S, Verhagen AP. Effect of routine diagnostic imaging for patients with musculoskeletal disorders: A meta-analysis. Eur J Intern Med. 2015 Oct;26(8):585-95. doi: 10.1016/j.ejim.2015.06.018. Epub 2015 Jul 15. PMID 26186812

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT07158892/Prot_SAP_000.pdf